CLINICAL TRIAL: NCT00891137
Title: A Phase I Trial to Determine Safety and Tolerability of Ex Vivo Expanded Human Myeloid Progenitor Cells (CLT-008) Infused 24 Hours Post-Transplant to Support Allogeneic Umbilical Cord Blood Transplantation for Hematologic Malignancies
Brief Title: Safety Study of Human Myeloid Progenitor Cells (CLT-008) After Cord Blood Transplant for Hematologic Malignancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cellerant Therapeutics (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MT 2008-38
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma; Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: adult acute myeloid leukemia 11q23 (MLL) abnormalities; adult acute myeloid leukemia inv(16)(p13;q22); adult acute myeloid leukemia t(15;17)(q22;q12); adult acute myeloid leukemia t(16;16)(p13;q22); adult acute myeloid leukemia t(8;21)(q22;q22); accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; childhood diffuse large cell lymphoma; childhood immunoblastic large cell lymphoma; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; extranodal marginal zone B-cell lymphoma; mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; stage I adult Burkitt lymphoma; contiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult Burkitt lymphoma; Waldenstrom macroglobulinemia; noncontiguous stage II adult immunoblastic; contiguous stage II adult immunoblastic; large cell lymphoma; stage I adult immunoblastic large cell lymphoma; previously treated myelodysplastic syndromes; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; refractory multiple myeloma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; splenic marginal zone lymphoma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; refractory anemia with excess blasts in transformation; refractory anemia with excess blasts; refractory anemia; prolymphocytic leukemia; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; refractory chronic lymphocytic leukemia; stage IV adult Burkitt lymphoma; stage I childhood small noncleaved cell lymphoma; stage II childhood small noncleaved cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage IV childhood small noncleaved cell lymphoma; recurrent childhood small noncleaved cell lymphoma; stage I childhood large cell lymphoma; stage II childhood large cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood large cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; stage I mantle cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; recurrent childhood large cell lymphoma; stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; recurrent childhood lymphoblastic lymphoma; childhood myelodysplastic syndromes; Burkitt lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Congenital Abnormalities; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Lymphoma, Large B-Cell, Diffuse; Leukemia, Myeloid, Chronic-Phase; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Waldenstrom Macroglobulinemia; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Anemia, Refractory, with Excess of Blasts; Anemia, Refractory; Leukemia, Prolymphocytic; Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Experimental): Low dose, single donor CLT-008 (human myeloid progenitor cells)
  Interventions: Biological: human myeloid progenitor cells
- Group B (Experimental): Low dose, multiple donor CLT-008 (human myeloid progenitor cells)
  Interventions: Biological: human myeloid progenitor cells
- Group C (Experimental): Intermediate dose, multiple donor CLT-008 (human myeloid progenitor cells)
  Interventions: Biological: human myeloid progenitor cells
- Group D (Experimental): High dose, multiple donor CLT-008 (human myeloid progenitor cells)
  Interventions: Biological: human myeloid progenitor cells

INTERVENTIONS:
Biological: human myeloid progenitor cells — Single intravenous injection/infusion
  Other Names: CLT-008; hMPC

SUMMARY:
Ex vivo expanded human myeloid progenitor cells (hMPCs; CLT-008) have the potential to accelerate neutrophil recovery in patients receiving myeloablative conditioning as part of an umbilical cord blood transplant for hematologic cancer. In this study, the safety and tolerability of CLT-008 administered 24 hours after an umbilical cord blood transplant will be determined by monitoring for adverse reactions, neutrophil and platelet recovery, hematopoietic chimerism, graft-versus-host disease (GVHD), and infections.

ELIGIBILITY:
Key Inclusion Criteria:

* Undergoing allogeneic (4-6/6 matched) umbilical cord blood graft with at least 2.5 x 10e7 cells/kg for hematological malignancy:

  * High risk acute myeloid leukemia (AML) in complete remission
  * Very high risk pediatric AML; patients <21 years eligible with <25% blasts in marrow after failed chemotherapy
  * High risk acute lymphocytic leukemia (ALL) in complete remission
  * Chronic myelogenous leukemia (CML), excluding refractory blast crisis
  * Myelodysplasia (MDS) IPPS Int-2 or high risk, or refractory anemia with severe pancytopenia or high risk cytogenetics
  * Chronic lymphocytic leukemia (CLL), small lymphocytic lymphoma (SLL), marginal zone B-cell lymphoma or follicular lymphoma that have progressed after two prior therapies
  * Lymphoplasmacytic, lymphoma, mantle-cell lymphoma, prolymphocytic leukemia after initial therapy and complete or partial remission
  * Large cell non-Hodgkin lymphoma (NHL) in second complete or partial remission (chemotherapy refractory large cell NHL not eligible)
  * Lymphoblastic lymphoma, peripheral T cell lymphoma including angioimmunoblastic lymphoma, Burkitt's lymphoma, and other high-grade NHL after initial therapy if stage III/IV in complete or partial remission, or after progression if stage I/II <1 year (chemotherapy refractory high-grade NHL not eligible)
  * Multiple myeloma beyond 2nd partial remission
* Preparative regimen consisting of cyclophosphamide, fludarabine, and total body irradiation
* Adequate organ function

Key Exclusion Criteria:

* Symptomatic underlying pulmonary disease or requiring oxygen
* Active infection
* HIV positive
* Pregnant or nursing

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 100 days post transplant

SECONDARY OUTCOMES:
Neutrophil and platelet recovery | 100 days post transplant
Persistence of CLT-008 derived cells | 100 days post transplant
Graft-versus-host disease (GVHD) | 100 days post transplant
Non-relapse mortality | 100 days post transplant
Infections | 42 days post transplant

CONTACTS AND LOCATIONS:
Overall Officials: John E Wagner, MD, Principal Investigator — University of Minnesota
Locations (8):
- United States (8):
  - Children's Hospital of Orange County, Orange, California
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Loyola University Medical Center, Cardinal Bernardin Cancer Center, Maywood, Illinois
  - University of Minnesota: Masonic Cancer Center, BMT Clinic, and Fairview Medical Center, Minneapolis, Minnesota
  - Cleveland Clinic, Taussig Cancer Institute, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: Cellerant Therapeutics, Inc. — http://www.cellerant.com